CLINICAL TRIAL: NCT06229938
Title: Detection of Hypovolemia in the Elderly Patient Undergoing Surgery
Acronym: HOOI
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Carolien SE Bulte, Principal investigator, Amsterdam UMC, location VUmc
Other Study IDs: ABR NL62141.029.17; METC 2018.009 (Other: Ethics Committee VUmc)
Record Dates: First submitted 2023-08-14; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Hypovolemia; Perioperative/Postoperative Complications
Keywords: Elderly
MeSH Terms: conditions — Hypovolemia; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly perioperative population: All patients included in the study (minimum 70 years of age on day of surgery)
  Interventions: Other: Passive leg raise manoeuvre

INTERVENTIONS:
Other: Passive leg raise manoeuvre — Stroke volume measurements are performed with the Nexfin hemodynamic monitor and the volemic state measurement is based on the principle of the classic passive leg raise test. The Nexfin monitor (Nexfin CC, Edwards Life Sciences, the Netherlands) uses a small inflatable cuff around the index finger of the right hand, to measure the blood pressure, and uses a specific algorithm to calculate the stroke volume.
  First a baseline measurement is performed during supine position while the patient is lying in bed. Next, the head end will be lowered until lying flat, and the legs will be passively raised until the lower end of the bed is 30 degrees elevated. The change in stroke volume following the passive leg raise test is used to assess fluid responsiveness. An increase of 10% indicates a fluid responsive status or hypovolemia.

SUMMARY:
Prospective observational study, in which the primary aim of the study is to determine the incidence of perioperative hypovolemia in the elderly patient scheduled for major surgery. Hypovolemia is defined as the presence of fluid responsiveness, which equals increase in stroke volume > 10% after a passive leg raise according to the Nexfin non-invasive cardiac output measurement.

This study aims to include 150 elderly patients aging 70 years or older undergoing scheduled major surgery. The passive leg raising test on 4 consecutive time points in the perioperative period.

DETAILED DESCRIPTION:
Rationale:

There is currently limited evidence available on the occurrence of perioperative hypovolemia in the elderly population, and whether this hypovolemic state is related to postoperative complications in these patients. More information regarding this relationship may be valuable in strategies aiming for a reduction in postoperative complications in the elderly. In particular, postoperative complications lead to long term morbidity, decrease quality of live, increase health care costs and are the most important factor of patient survival. Therefore, the present study aims to investigate how many elderly patients suffer from hypovolemia in the perioperative period, and how this relates to postoperative complications.

Objective:

The primary aim of the study is to determine the incidence of perioperative hypovolemia in the elderly patient scheduled for major surgery. Hypovolemia is defined as the presence of fluid responsiveness, which equals increase in stroke volume > 10% after a passive leg raise according to the Nexfin non-invasive cardiac output measurement.

Study design:

Open, prospective, observational study

Study population:

150 elderly patients aging 70 years or older undergoing scheduled major surgery.

Intervention:

Passive leg raising test on 4 consecutive time points in the perioperative period

Main study endpoints:

Relative number of patients that have a change in stroke volume of more than 10% upon a passive leg raising test.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

One of the investigators will visit the ward and will use the inflatable blood pressure cuff around the index finger of the right hand. The measurement will be performed while sitting and is continued for 5 minutes after lowering the head end of the bed and raising the lower end of the bed. As the bed functions electronical the change in movement occurs slowly and without any effort. Overall discomfort associated with these tests is regarded to as minimal. There are no benefits related to participation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 70 years or older
* Scheduled for elective surgery
* Procedures with expected postoperative stay of at least two days

Exclusion Criteria:

* Procedure in ambulatory practice
* Acute surgery
* Patients with current cardiac arrhythmias
* Symptoms of cardiovascular shock or decompensation at presentation
* Impossible to perform measurements due to patient characteristics
* Inability to comprehend patient information and consequences of the study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 150 elderly patients aging 70 years or older admitted to the hospital for scheduled major surgery. Major surgery will be defined as an expected length of stay being at least two postoperative days as these carry the greatest complication risk, including gastro-intestinal, pulmonary, major gynecological or urological and vascular surgery.
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Incidence of hypovolemia (%) | Preoperatively; and postoperatively (at 2, 24 and 48 hours postoperatively)
  preoperative incidence of hypovolemia (stroke volume increase of 10% or more upon a passive leg raising manoeuvre)

SECONDARY OUTCOMES:
Postoperative complications | 30 day
  All complications (descriptive); classified conform Clavien-Dindo classification
Postoperative mortality | 30 day
  mortality
Postoperative care | 30 day
  Unplanned Intensive Care Unit admission (categorical: yes/no); and if applicable for how long (continuous; in days).
Blood transfusion | intra-operative (duration of surgical procedure)
  Erythrocytes concentrate transfusion (continuous scale; number of units)
Fluid administration | intra-operative (duration of surgical procedure)
  All fluids administered: including crystalloids, colloids, medication, all blood product (continuous scale, in mL)
Vaso-active therapy | intra-operative (duration of surgical procedure)
  Use of vaso active medication, including norepinephrine; epinephrine; dobutamine; atropine; phenylephrine; ephedrine (categorical: yes/no).
Duration of surgery | intra-operative (duration of surgical procedure)
  Duration of surgical procedure (continuous scale; in minutes)
Anesthetic technique | intra-operative (duration of surgical procedure)
  Type of anesthesia (nominal categories; general anesthesia; spinal; epidural; or mixed)

CONTACTS AND LOCATIONS:
Overall Officials: Carolien Bulte, Phd, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No